CLINICAL TRIAL: NCT06781177
Title: Comparison of Total Intravenous Anesthesia Methods in Terms of Postoperative Outcomes in Thoracolumbar Spinal Surgery Cases
Brief Title: Comparison of Total Intravenous Anesthesia Methods in Spinal Surgery (TIVA)
Acronym: TIVA
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aysegul Danaci, specialist doctor, anesthesiologist, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2023-05/204
Record Dates: First submitted 2024-12-29; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia
Keywords: Anesthesia, Intravenous; Bispectral Index Monitor; Ketamine; Lidocaine; Spinal Fusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group S: Propofol at 30-100 mcg/kg/min and remifentanil at 0.05-0.2 mcg/kg/min (classical TIVA)
- Group K: Propofol at 30-100 mcg/kg/min, remifentanil at 0.05-0.1 mcg/kg/min, ketamine at 5 mcg/kg/min
- Group L: Propofol at 30-100 mcg/kg/min, remifentanil at 0.05-0.1 mcg/kg/min, lidocaine at 1.2 mg/kg/h

SUMMARY:
This study aims to compare the effects of the classical Total Intravenous Anesthesia (TIVA) method and multimodal anesthesia protocols created by adding lidocaine and ketamine infusions on postoperative pain management, opioid consumption, and surgical recovery in posterior thoracolumbar spinal fusion surgeries.

A prospective observational study was conducted with 72 patients undergoing posterior thoracolumbar spinal fusion surgeries. Patients were evenly divided into three groups: classical TIVA (propofol and remifentanil), TIVA + ketamine, and TIVA + lidocaine. Hemodynamic parameters and drug dosages were recorded during the intraoperative period, while pain scores, opioid consumption, time to first ambulation and bowel movement, as well as nausea-vomiting and sedation scores, were documented postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* ASA classification I-III
* Patients undergoing posterior thoracolumbar spinal surgery and neuromonitoring under general anesthesia

Exclusion Criteria:

* Emergency operations
* Pregnant patients
* Patients with ASA classification IV or higher*
* Patients allergic to morphine and local anesthetics
* Patients with neurological or psychiatric disorders (on ongoing antidepressant and/or anticonvulsant therapy) Illiterate patients
* Patients unable to cooperate
* Extremely low or high body weight (less than 40 kg or more than 100 kg)
* Chronic opioid use
* Diabetes mellitus (DM) requiring insulin therapy
* Chronic alcohol use
* Patients with peripheral neuropathy
* Patients with cardiac arrhythmias

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older, classified as ASA I-III, undergoing posterior thoracolumbar spinal surgery and neuromonitoring under general anesthesia, and fluent in Turkish.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score Using Visual Analog Scale (VAS) | postoperative 24 hours
  Pain levels will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain), at 30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours postoperatively.
Total Opioid Consumption in the First 24 Hours Postoperatively | Postoperative 24 hours
  The total amount of opioids administered during the first 24 hours postoperatively will be recorded and converted to morphine milligram equivalents (MME).

SECONDARY OUTCOMES:
Time to First Ambulation After Surgery | postoperative 24 hours
  The time from the end of surgery to the patient's first ambulation will be recorded in hours.
Time to First Bowel Movement After Surgery | postoperative 24 hours
  The time from the end of surgery to the patient's first reported bowel movement will be recorded in hours.
Incidence of Nausea and Vomiting | postoperative 24 hours
  The presence of postoperative nausea and vomiting will be recorded within the first 24 hours after surgery.
Opioid Requirement Within After Surgery | postoperative 1 month
  The need for opioid use within 1 month after discharge will be evaluated through follow-up phone calls. The percentage of patients requiring opioids during this period will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Abdurrahman Yurtaslan Oncology Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

DOCUMENTS (3):
  • Study Protocol (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT06781177/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT06781177/SAP_001.pdf
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT06781177/ICF_002.pdf